CLINICAL TRIAL: NCT03278587
Title: Village-Integrated Eye Worker Trial II - Pilot
Acronym: VIEW II Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Seva Foundation (Other); Bharatpur Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-22776
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Cataract; Glaucoma; Age Related Macular Degeneration; Diabetic Retinopathy; Refractive Errors
MeSH Terms: conditions — Cataract; Glaucoma; Macular Degeneration; Diabetic Retinopathy; Refractive Errors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Community-based screening (Active Comparator)
  Interventions: Other: Community-based screening program
- Cataract camp program (Active Comparator)
  Interventions: Other: Cataract camp program
- Community health worker program (Active Comparator)
  Interventions: Other: Community health worker program
- No intervention (No Intervention)

INTERVENTIONS:
Other: Community-based screening program — In communities randomized to receive the screening program, all adults aged 50 and older will be eligible to receive screening for ocular disease. Screening assessments include visual acuity, refraction, intra-ocular pressure, fundus photography, and anterior segment photography. Participants meeting criteria for referral based on screening assessments will be referred to the nearest eye care center or eye hospital for further evaluation.
  Arms: Community-based screening
Other: Cataract camp program — In communities randomized to receive the cataract camp program, all adults aged 50 and older will be eligible to participate in a routine cataract camp run by Bharatpur Eye Hospital. Trained ophthalmic personnel and assistants will perform case detection for cataract via visual acuity, pen light exam, and indirect ophthalmoscope exam per Bharatpur Eye Hospital's standard cataract camp program. Participants with cataracts will be referred to the nearest eye care center or eye hospital for further evaluation.
  Arms: Cataract camp program
Other: Community health worker program — In communities randomized to receive the community health worker program, all adults aged 50 and older will be eligible to participate. Existing community health workers will be trained to perform case detection for cataract via visual acuity assessment. Participants with cataracts will be referred to the nearest eye care center or eye hospital for further evaluation.
  Arms: Community health worker program

SUMMARY:
The vast majority of blindness is avoidable. The World Health Organization (WHO) estimates that 80% of cases of visual impairment could be prevented or reversed with early diagnosis and treatment. The leading causes of visual impairment are cataract and refractive error, followed by glaucoma, age-related macular degeneration (AMD), and diabetic retinopathy (DR). Loss of vision from these conditions is not inevitable; however, identifying at-risk cases and linking cases with appropriate care remain significant challenges.

Worldwide, eye health care systems must determine optimal strategies for reaching people outside of their immediate orbit in order to reduce visual impairment. Visual impairment can be reduced by case detection of prevalent disease like cataract and refractive error, or by screening for early disease like glaucoma, AMD, and DR and preventing progression. Systems around the world have developed numerous approaches to both case detection and screening but there is very little research to support the choice of allocating resources to case detection or screening and little data exists on the cost effectiveness of the various approaches to each.

VIEW II Pilot is a cluster-randomized trial to determine the effectiveness of different approaches to community-based case detection and screening for ocular disease. Communities in Nepal will be randomized to one of four arms: 1) a comprehensive ocular screening program, 2) a cataract camp-based program, 3) a community health worker-based program, and 4) no program.

DETAILED DESCRIPTION:
Specific Aim 1: to determine whether screening leads to increased visual acuity compared to the cataract camp approach.

Specific Aim 2: to determine whether a community health volunteer program increases the rate of cataract surgery compared to a no program.

ELIGIBILITY:
Inclusion Criteria(community-level):

* Wards in the Chitwan and Nawalparasi districts that participated in the VIEW trial and have not received a cataract camp in the past 6 months.

Inclusion Criteria (individual-level):

* Individuals aged 50 and older will be eligible to participate in the screening program, cataract camp programs, and the FCHV program

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16075 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 1 year
  Primary outcome for specific aim 1, comparison between screening and case detection arms
Cataract surgical rate | 1 year
  Primary outcome for specific aim 2, comparison between community health worker program and no program arms

SECONDARY OUTCOMES:
Cost-effectiveness | 1 year
  Cost-effectiveness of all 4 arms will be assessed
Visual acuity | 1 year
  Visual acuity of population 50 years and older in all arms will be compared
Number of cases of ocular disease detected | 1 year
  Number of cases of ocular disease in the screening and case detection arms will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Keenan, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Bharatpur Eye Hospital, Bharatpur, Chitwan, Nepal